CLINICAL TRIAL: NCT07346989
Title: Effectiveness of Non-invasive Brain Stimulation on Functional Capacity in Prefrail Older Adults
Brief Title: Non-invasive Brain Stimulation on Functional Capacity in Prefrail Older Adults
Acronym: NeuroFit
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Marta Inglés de la Torre, Professor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025-FIS-4007899
Record Dates: First submitted 2025-12-03; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Prefrail Elderly
Keywords: Prefrail; Non-invasive neuromodulation; TMS; TDCS; Virtual running; Functional capacity; Elderly
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- rTMS group (Experimental)
  Interventions: Other: rTMS
- rTMS placebo group (Placebo Comparator)
  Interventions: Other: rTMS placebo
- tDCS group (Experimental)
  Interventions: Other: tDCS
- tDCS placebo group (Placebo Comparator)
  Interventions: Other: tDCS placebo
- VR group (Experimental)
  Interventions: Other: Virtual running
- VR placebo group (Placebo Comparator)
  Interventions: Other: Virtual running placebo

INTERVENTIONS:
Other: rTMS — 24 HF-TMS sessions, 3 per week, with a duration of 20 minutes. Magnetic stimulation will be applied using a Neuro-MS/D transcranial magnetic stimulator (Neurosoft ®, Ivanovo, Russia) with a figure-eight coil. The coil will be placed tangentially to the skull in an anteromedial direction at 45º of M1 in the left hemisphere.
  They will then carry out a therapeutic exercise protocol (common to all groups) that will consist of performing lower limb exercises, including coordination, strength, balance and stretching exercises. The Borg Scale will be used to measure each person's perception of their effort, dyspnea and fatigue during each physical exercise.
  Arms: rTMS group
Other: rTMS placebo — The instrumentation will be the same as in the intervention with real rTMS, but the device will not emit any type of electrical stimulus. They will then perform the therapeutic exercise protocol explained above
  Arms: rTMS placebo group
Other: tDCS — The tDCS will be performed anodically (a-tDCS), and for 24 sessions, 3 days a week. The electrodes will be mounted on a neoprene helmet, in accordance with the International Standard 10-20 EEG System, for optimal targeting of the primary motor cortex M1. It will be a type of unihemispheric application, in which the anode will be located in the primary motor cortex (M1), and the cathode located in the orbitofrontal cortex contralateral to the anode. The treatment parameters will be: stimulation time of 20 minutes; intensity of 2mA, current rise-fall time at the beginning and end of stimulation of 30 seconds. They will then perform the therapeutic exercise protocol explained above.
  Arms: tDCS group
Other: tDCS placebo — The instrumentation will be the same as in the actual tDCS intervention, but the device will be programmed to increase the intensity from 0 to 2 mA progressively during the first 30 seconds and then cease to provide the patient with the initial itchy sensation on the skin, similar to the real application. They will then perform the therapeutic exercise protocol explained above.
  Arms: tDCS placebo group
Other: Virtual running — 24 sessions will be applied, 3 days a week. The patient will be placed standing (with an ad-hoc designed assistance system) in front of a mirror (located at waist height) and a height-adjustable screen (from waist to caudal) where a video of real legs running on a treadmill will be projected. In order for the participant to feel the projected legs as their own, people with different body sizes will have been previously recorded running to have recordings with legs of different size and length. Each session will last 20 minutes. They will then perform the therapeutic exercise protocol explained above.
  Arms: VR group
Other: Virtual running placebo — The instrumentation of the participants will be the same as in the intervention with virtual running. However, the projection will consist of a series of videos of landscapes in which no type of human or animal movement will appear in order not to stimulate the motor areas of the brain. They will then perform the therapeutic exercise protocol explained above.
  Arms: VR placebo group

SUMMARY:
The general objective of this study is to evaluate the effectiveness of non-invasive neuromodulation combined with a therapeutic exercise program on neuroplasticity and, therefore, on variables related to functional capacity and quality of life, in prefrail older adults.

DETAILED DESCRIPTION:
Three non-invasive neuromodulation strategies (Virtual Running, Transcranial Magnetic Stimulation (TMS) and Transcranial Direct Current Stimulation (tDCS)) will be studied. Thus, 3 sub-studies will be carried out (one for each intervention) and a comparison of the three interventions will be made, as described in the following sections. As specific objectives, for each of these sub-studies, the effect of the intervention program will be analyzed on: gait speed, general physical condition, frailty condition, static and dynamic functionality and gait quality, upper limb and lower limb isometric strength, quality of life, and neuroplasticity, in terms of plasma BDNF levels, in prefrail older adults.

ELIGIBILITY:
Inclusion Criteria:

* Age between 65 -90 years old
* Meet 1-2 frailty criteria, according to Fried's Criteria.
* Ability to understand instructions (Mini-Mental State Examination >23 points).
* Signing of the informed consent.

Exclusion Criteria:

* History of stroke within the past 6 months or hospital admission for any reason within the past 3 months.
* Alterations of the central or peripheral nervous system
* Alterations of the vestibular system
* Concomitant diseases
* Have a neurological pathology, cardiovascular musculoskeletal that contraindicates physical activity
* Epilepsy or history, medications that lower the seizure threshold
* Cardiac pacemaker, endocranial and hearing implants
* History of severe headaches
* Uncontrolled intracranial or arterial hypertension
* Heart and/or respiratory failure
* Implanted medication pump
* Skin lesions (psoriasis, eczema)
* Serious head surgeries
* Completing less than 80% of training sessions

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Frailty Condition | Five assessments: Baseline (T1); After the first session, at Day 1 (T2); Mid-term assessment, 4 weeks after the intervention starts (T3); After the intervention, 8 weeks (T4); Four weeks after the end of the intervention (follow-up assessment) (T5).
  Fried's criteria (Frailty Phenotype) will be used. Briefly, the participant will be considered frail if he or she meets three or more of the following criteria: i) unintentional weight loss greater than 4.5 kg in the last year; ii) feeling of general exhaustion, reported by the patient himself; iii) low level of physical activity; (iv) slowness of progress; v) muscle weakness, assessed by handgrip strength. Those patients who meet one or two criteria will be considered pre-frail and those who do not meet either will be considered non-frail
Walking speed | Five assessments: Baseline (T1); After the first session, at Day 1 (T2); Mid-term assessment, 4 weeks after the intervention starts (T3); After the intervention, 8 weeks (T4); Four weeks after the end of the intervention (follow-up assessment) (T5).
  The 10m Walking Test will be used to assess the speed of the walk, which records the time needed to cover the distance of 10m. The higher the walking speed, the greater the functional capacity

SECONDARY OUTCOMES:
Neuroplasticity | Three assessments: Baseline (T1); After the intervention, 8 weeks (T4); Four weeks after the end of the intervention (follow-up assessment) (T5).
  Neruoplasticity will be determined from the concentration of BDNF in plasma. A nurse will draw blood samples in BD Vacutainer® tubes, with EDTA as an anticoagulant. It will be centrifuged at 1500 G for 15 minutes at 4⁰ C, the supernatant (plasma) will be collected in eppendorf type tubes, which will be frozen at -80⁰ C until subsequent analysis. For the determination of BDNF levels, the ChemiKine™ BDNF Sandwich kit for ELISA (Millipore, Temecula, CA, USA) will be used, according to the manufacturer's instructions
Heart rate variability | Five assessments: Baseline (T1); After the first session, at Day 1 (T2); Mid-term assessment, 4 weeks after the intervention starts (T3); After the intervention, 8 weeks (T4); Four weeks after the end of the intervention (follow-up assessment) (T5).
  HRV will be measured during 5 minutes at rest before intervention and during 20 minutes while performing aerobic exercise (walking). HRV will be measured with the PolarH10 band (Polar ®, Finland).
Muscle strength | Three assessments: Baseline (T1); After the intervention, 8 weeks (T4); Four weeks after the end of the intervention (follow-up assessment) (T5).
  Measurement of the isometric action of the lower limb muscles will be carried out by means of a load cell (Chronojump, Spain) connected to the corresponding software (Chronojump Boscosystem). Specifically, the isometric strength of the gluteus medius, quadriceps, and hamstrings will be measured. The participant will be asked for a maximum of three repetitions with a duration of five seconds each, and a rest between them of another thirty seconds. The maximum value will be recorded, as well as the average value of each of the three repetitions, and the average will then be obtained, which will be the variable used for the subsequent data analysis. As for upper limb strength, assessed by grip strength, this will be determined by a Lafayette hand dynamometer. 3 measurements of the dominant hand will be taken and the mean will be taken for further analysis. Higher values indicate greater muscle strength
Quality of life EQ-5D | Three assessments: Baseline (T1); After the intervention, 8 weeks (T4); Four weeks after the end of the intervention (follow-up assessment) (T5).
  Determined using the EQ-5D instrument, a measure of self-perceived health, consisting of two parts: the EQ-5D descriptive system, which assesses five dimensions of health (i.e. mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) and a visual analogue scale (VAS), in which people must estimate their general health status on a scale from 0 to 100. Higher values indicate greater quality of life.
Lower limb muscle power | Five assessments: Baseline (T1); After the first session, at Day 1 (T2); Mid-term assessment, 4 weeks after the intervention starts (T3); After the intervention, 8 weeks (T4); Four weeks after the end of the intervention (follow-up assessment) (T5).
  It will be recorded with the 5 times sit to stand test (5STST). The participant must sit down and get up from a chair and the time it takes to perform the activity is timed. The higher the speed, the greater lower limb power
Static and dynamic functionality and gait quality | Five assessments: Baseline (T1); After the first session, at Day 1 (T2); Mid-term assessment, 4 weeks after the intervention starts (T3); After the intervention, 8 weeks (T4); Four weeks after the end of the intervention (follow-up assessment) (T5).
  For this assessment, the FallSkip® tool will be used, which allows, by means of an inertial sensor incorporated in a smartphone, to record variables such as the medium-lateral and vertical displacement of the center of pressures in both dynamic and static, as well as to record the power to sit and get up from a chair and the variability of movement in a modified protocol of the Timed up and Go test. Based on the calculation of these variables, FallSkip® provides a fall risk score for each patient, ranging from very low, low, moderate, high, to very high risk, depending on the results obtained during the different test phases.
Static and dynamic functionality and gait quality with a dual task | Three assessments: Baseline (T1); After the intervention, 8 weeks (T4); Four weeks after the end of the intervention (follow-up assessment) (T5).
  For this assessment, the FallSkip® tool will be used, which allows, by means of an inertial sensor incorporated in a smartphone, to record variables such as the medium-lateral and vertical displacement of the center of pressures in both dynamic and static, as well as to record the power to sit and get up from a chair and the variability of movement in a modified protocol of the Timed up and Go test. Based on the calculation of these variables, FallSkip® provides a fall risk score for each patient, ranging from very low, low, moderate, high, to very high risk, depending on the results obtained during the different test phases. For the dual task, a simultaneous activity will be used that will consist of numerical subtraction while walking. The higher punctuation, the better dual task functionality.

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared under request to the authors

REFERENCES:
- [Background] Molla-Casanova S, Page A, Lopez-Pascual J, Ingles M, Sempere-Rubio N, Aguilar-Rodriguez M, Munoz-Gomez E, Serra-Ano P. Effects of mirror neuron activation therapies on functionality in older adults: Systematic review and meta-analysis. Geriatr Nurs. 2024 Mar-Apr;56:115-123. doi: 10.1016/j.gerinurse.2024.02.006. Epub 2024 Feb 11. PMID 38346365
- [Background] Global Recommendations on Physical Activity for Health. Geneva: World Health Organization; 2010. Available from http://www.ncbi.nlm.nih.gov/books/NBK305057/ PMID 26180873
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156